CLINICAL TRIAL: NCT06625892
Title: Investigating the Related Factors and Outcome of Kinesiophobia and the Effects of Multidimensional Interventions in Cardiac Surgery Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ai-Ling Chang (Other)
Collaborators: Da-Yeh University (Other)
Responsible Party: Sponsor-Investigator, Ai-Ling Chang, Supervisor, Changhua Christian Hospital
Organization: Changhua Christian Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 231124
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Diseases Requiring Surgery
Keywords: kinesiophobia, cardiac surgery
MeSH Terms: conditions — Kinesiophobia

STUDY DESIGN:
Intervention Model Description: The first-year research adopts a descriptive, correlational, and repeated-measures design, while the second-year research employs an experimental design. Participants are randomly assigned to either the experimental or control group. The experimental group undergoes a 12-week comprehensive intervention, while the control group receives no intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessors dose not know the allocation of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- the interventions group (Experimental): The experimental group undergoes a 12-week multidimensional interventions.
  Interventions: Behavioral: the multidimensional interventions
- the control group (No Intervention): the control group receives no intervention.

INTERVENTIONS:
Behavioral: the multidimensional interventions — The study participants will receive cognitive behavior therapy intervention for six weeks, one session per week, 45 minutes each time, and exercise training for twelve weeks, twice sessions per week, 60 minutes each time.
  Arms: the interventions group

SUMMARY:
The primary objective of this two-year research project is to investigate the status of activity fear, its related factors, and prognosis in cardiac surgery patients in the first year. Subsequently, the study aims to develop a comprehensive intervention strategy combining exercise with cognitive-behavioral approaches tailored for cardiac surgery patients and assess the effectiveness of this intervention on activity fear, prognosis, and quality of life in the second year.

DETAILED DESCRIPTION:
The study uses a convenient sampling method, focusing on patients undergoing cardiac surgery in the cardiac surgery ward of the Central Medical Center. The first-year research adopts a descriptive, correlational, and repeated-measures design, while the second-year research employs an experimental design. Participants are randomly assigned to either the experimental or control group. The experimental group undergoes a 12-week multidimensional interventions, while the control group receives no intervention. Data are collected through structured questionnaires. Data collection occurs at discharge, two weeks post-discharge, six weeks, 12 weeks, and 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients received cardiac surgery.
* Aged 18 or above.
* Clear consciousness and able to communicate in Mandarin or Taiwanese.
* Willing and consent to participate after being informed of the study purpose and procedures.

Exclusion Criteria:

* Cognitive impairment,
* Psychiatric disorders, and
* Long-term bedridden patients who rely on others for daily activities.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 245 (Estimated)
Dates: Start 2024-08-14 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
kinesiophobia | 1 day discharge, two weeks post-discharge, six weeks, 12 weeks, and 24 weeks.
  Tampa Scale of Kinesiophobia for Heart (TSK Heart) was used for measuring kinesiophobia in this study. The TSK Heart developed by Bäck et al. (2012), assesses fear of movement in patients with coronary artery disease. It comprises four dimensions: exercise avoidance, fear of injury, dysfunctional self-perception, and perceived risk of heart problems, with 17 items. Each item is scored on a 4-point Likert scale (1 = strongly disagree to 4 = strongly agree), and items 4, 8, 12, and 16 are reverse scored. The total score ranges from 17 to 68, with higher scores indicating greater fear of movement. A TSK Heart score below 37 indicates a low fear of movement, while a score of 37 or higher indicates a high fear of movement. The scale's intra-class correlation coefficient is 0.83, and its internal consistency (Cronbach's alpha) is 0.78 (Bäck et al., 2012).

SECONDARY OUTCOMES:
International Physical Activity Questionnaire (IPAQ) | 1 day discharge, two weeks post-discharge, six weeks, 12 weeks, and 24 weeks.
  This study uses the short form of the Taiwan version of the IPAQ, developed in collaboration with Liu Ying-Mei and the World Health Organization. It consists of 7 items assessing physical activity over the past week across work, household chores, transportation, and leisure activities, including time and frequency of walking, moderate and vigorous activities, and time spent sitting. The total physical activity is calculated by multiplying each activity category by its corresponding Metabolic Equivalent (MET), execution time, and activity days. An IPAQ score below 600 indicates low physical activity, 600-3000 indicates moderate physical activity, and above 3000 indicates high physical activity. The scale's content validity is 0.994, and its intra-class correlation coefficient is 0.704 (Liou et al., 2008).
Taiwan Brief Version of the World Health Organization Quality of Life Questionnaire (WHOQOL-BREF) | 1 day discharge, two weeks post-discharge, six weeks, 12 weeks, and 24 weeks.
  Professor Yao Kai-Ping developed this questionnaire after obtaining authorization; this questionnaire assesses the quality of life across four domains: physical health, psychological well-being, social relationships, and environment, with 28 items. Each item is scored on a 5-point scale. Scores for each domain are calculated by averaging the scores of the items within that domain and multiplying by 4. Items 3, 4, and 26 are reverse-scored by subtracting the original score from 6. Higher scores indicate a better quality of life. The internal consistency is 0.91, and the content validity of the domains ranges from 0.51 to 0.64 (Taiwan WHOQOL Group, 2000; Yao Kai-Ping, 2002).

CONTACTS AND LOCATIONS:
Overall Officials: Wan-Ting Huang, PhD, Principal Investigator — Da-Yeh University
Locations (1):
- Changhua Christian Hospital, Changhua, Taiwan